CLINICAL TRIAL: NCT02872571
Title: Evaluation of the Efficacy of Intramuscular Islet Autograft After Extensive Pancreatectomy
Acronym: AUTOGRAFTIM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010_49; 2012-A00312-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2020-09

CONDITIONS: Disorder of Endocrine Pancreas
Keywords: islet of Langerhans; transplantation; muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intramuscular Islet Autograft (Experimental): Intramuscular Islet Autograft After Extensive Pancreatectomy
  Interventions: Drug: Intramuscular Islet Autograft

INTERVENTIONS:
Drug: Intramuscular Islet Autograft — Intramuscular Islet Autograft After Extensive Pancreatectomy

SUMMARY:
The liver may not be an optimal site for islet transplantation due to obstacles by an instant blood-mediated inflammatory response, and low revascularization of transplanted islets. Therefore, intramuscular islet transplantation offers an attractive alternative, based on its simplicity, enabling easier access for noninvasive graft imaging and cell explantation.

DETAILED DESCRIPTION:
The field of β cell replacement therapies has progressed extensively over the last decades. It is well established that successful intraportal islet transplantation can restore endogenous β cell function to subjects with type 1 diabetes mellitus. In fact, when the graft function is optimal, insulin independence can be consistently prolonged for up to 5 years in 50% of patients. Several factors influence the outcome and performance of the graft upon implantation. For instance, preclinical studies have confirmed the significant differences in utilizing several sites for the implantation of islet grafts, but the most utilized clinical approach is embolization into the liver. However, it has become evidently clear that the liver may not be the optimal environment as a recipient site for pancreatic islets, owing not only to immunologic, but also to anatomic and physiologic factors that may promote a decline in islet function. Moreover, intrahepatic islet infusion is often associated with an immediate blood- mediated inflammatory reaction , thrombosis and hepatic tissue ischemia with elevated blood liver enzymes. In addition, the cross-talk between activated coagulation and inflammatory mediators after implantation, dramatically affects islet cell survival and engraftment, resulting in β cell dysfunction or death, depicting primary nonfunction as a consequence of reduced functional islet mass. This intrahepatic environment appears to potently impair the metabolic functions of transplanted islets. Furthermore, the complications associated with graft recovery within the hepatic site, will further limit its potential applications in exploiting insulin-secreting cells obtained from alternative cell sources. These include xenogenic islets, immortalized β cell lines, embryonic stem cells, or adult progenitor cells, including β cell encapsulation.

Restoration of β cell function is a highly desirable goal for patients with unstable diabetes; therefore, the search for an alternative site that is safer for islet transplantation is imperative.

In man, autotransplantation of minced tissue into striated muscle following blunt dissection has been successfully used in parathyroid surgery for several decades. Initially demonstrated in rodents in the early 1980s, intramuscular islet transplantation (IMIT) has rarely been considered as a clinically feasible implantation site.

This study want to provide direct evidence of the feasibility and function of autologous islets transplanted in the muscle

ELIGIBILITY:
Inclusion Criteria:

age over 18 years indication for pancreatectomy for benign pancreatic disease not genetically determined (chronic pancreatitis, ductal lesions, neuroendocrine or cystic tumors) or pancreatic trauma

Exclusion Criteria:

Patients with suspected lesion genetically determined or malignant on the basis of preoperative and / or during surgical exploration and / or during pathological examination Refusal to sign the consent form Patient not affiliated with a social security scheme Pregnant or lactating women Persons deprived of liberty, person under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients with a functioning graft in the arm 3 months after autograft. | 3 months
  Graft function will be estimated by the difference in insulin response between the two arms after the test stimulus by arginine (Acute Insulin Response or AIRarg) .The graft will be considered functional (success) when the insulin response in the grafted arm will be at least 30% higher compared to the other arm, 3 months after transplantation.

SECONDARY OUTCOMES:
The percentage of patients with a functioning graft in the arm | 6 months, 12 months
  To demonstrate the function of transplanted islets in the arm in patients receiving autologous islet intramuscularly after undergoing pancreatectomy for benign lesion extent, to prevent post surgical diabetes.
Continuous Glucose Monitoring System | at baseline ( before autograft) at 3,6,12 months
  Continuous recording of blood glucose during 72 hours by Continuous Glucose Monitoring System
Oral Glucose Tolerance Test | at baseline ( before autograft) at 3,6,12 months
  The glucose tolerance test is a medical test in which glucose is given and blood samples taken afterward to determine how quickly it is cleared from the blood.
hemoglobin A1c (HbA1c) blood test | at baseline ( before autograft) at 3,6,12 months
  HbA1c measures blood glucose levels over a period of time.

CONTACTS AND LOCATIONS:
Overall Officials: François Pattou, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - Chu Amiens Picardie, Amiens
  - CHRU, Hôpital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No